CLINICAL TRIAL: NCT05918107
Title: Phase II Clinical Trial to Evaluate the Preliminary Efficacy, Safety and Pharmacokinetic Characteristics of PM8002 Injection Combined With Standard Chemotherapy in the First-line Treatment of Subjects With Inoperable Malignant Mesothelioma
Brief Title: A Study of PM8002 Injection in Combination With Standard Chemotherapy as First Line Therapy in MPM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM8002 -B003C-MPM-R
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: MPM
Keywords: First line
MeSH Terms: interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002+pemetrexed+platinum (Other): Subjects will be administered with PM8002 plus pemetrexed+platinum via intravenously (IV) Q3W for 4-6 cycles,followed by PM8002 until disease progression intolerable toxicity for a maximum of 2 years.
  Interventions: Drug: PM8002; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: PM8002 — IV infusion
Drug: Pemetrexed — IV infusion
Drug: Cisplatin — IV infusion
Drug: Carboplatin — IV infusion

SUMMARY:
PM8002 is a bispecific antibody targeting PD-L1 and VEGF. This study will evaluate the efficacy and safety of PM8002 in combination with pemetrexed and platinum as first line treatment for MPM.

DETAILED DESCRIPTION:
PD-L1 and VEGF play important roles in immune escape and tumor angiogenesis and enhance cancer growth and metastasis. PM8002 is a bispecific antibody targeting PD-L1 and VEGF-A. Here, the investigators present the results from a Phase II study of PM8002 in combination with pemetrexed and platinum subjects in unresectable malignant mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in clinical research; fully understand the study and voluntarily sign the informed consent; willing to follow and have the ability to complete all trial procedures;
2. Male or female, aged ≥18 years;
3. Malignant mesothelioma confirmed by histology, without indication for surgery;
4. Have not received systemic anti-tumor therapy in the past (if the subject has received neoadjuvant or adjuvant chemotherapy in the past, the last treatment time must be more than 6 months from the time of recurrence);
5. Sufficient organ function;
6. Eastern Cooperative Oncology Group (ECOG) physical status (PS) score is 0-1;
7. Expected survival period ≥ 12 weeks;
8. There is at least one measurable lesion (malignant pleural mesothelioma is based on mRECIST version 1.1, and malignant mesothelioma in other parts is based on RECIST version 1.1).

Exclusion Criteria:

1. History of severe allergic diseases, severe drug (including unmarked test drug) allergy history, or known allergy to any component of the drug in this study;
2. Brain parenchymal metastases or meningeal metastases with clinical symptoms, judged by the investigators as not suitable for inclusion;
3. Had other active malignant tumors within 5 years before starting the study drug treatment, except for malignant tumors that can be treated locally and cured (such as skin basal cell or squamous cell carcinoma, superficial or non-invasive bladder cancer), cervical carcinoma in situ, breast ductal carcinoma in situ, papillary thyroid carcinoma);
4. Currently there are uncontrollable pleural, pericardial, and peritoneal effusions, and those with catheter drainage also need to be excluded;
5. Unexplained fever > 38.5°C before starting the study treatment (judged by the investigator, fever caused by tumor can be included in the group);
6. There is uncontrollable tumor-related pain, and those who need analgesic treatment should have a stable analgesic treatment plan at the time of screening; asymptomatic metastatic lesions, if they grow further, may cause dysfunction or intractable pain (such as current and spinal cord compression unrelated epidural metastases), local therapy should be considered before screening if appropriate;
7. Currently have clear interstitial lung disease or non-infectious pneumonia, except radiation pneumonitis caused by local radiotherapy;
8. There are active infections;
9. Have a history of immunodeficiency, including a positive test for human immunodeficiency virus (HIV) antibodies;
10. Positive for syphilis antibody;
11. Expect to receive any other forms of anti-tumor drug treatment during the trial period;
12. Those who have received allogeneic hematopoietic stem cell transplantation or organ transplantation in the past;
13. Pregnant or lactating women;
14. According to the investigator's judgment, the subject's basic condition may increase the risk of receiving the study drug treatment, or cause confusion for the explanation of the toxic reaction and AE;
15. Other investigators think that they are not suitable to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-08-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | : Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment]
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Duration of response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Progression free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Jilin Provice Cancer Hospital
Locations (1):
- Jilin Provincial Tumor Hospital, Changchun, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations.
Time Frame: After the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy